CLINICAL TRIAL: NCT02958033
Title: Shandong Cancer Hospital Affiliated to Shandong University
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Min Xu, Principal Investigator, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shandong Cancer Hospital
Record Dates: First submitted 2016-10-18; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Early-stage Breast Cancer; Breast Conserving Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HF WBI-SIB breast radiation (Experimental): WBI-SIB breast radiation(WBI 2.5Gy x18 and SIB 2.88Gy x18)
  Interventions: Radiation: Whole Breast irradiation Plus simultaneous tumor bed Boost
- CF WBI-SIB breast radiation (Placebo Comparator): WBI-SIB breast radiation(WBI 1.8Gy x28 and SIB 2.15Gy x28)
  Interventions: Radiation: Whole Breast irradiation Plus simultaneous tumor bed Boost

INTERVENTIONS:
Radiation: Whole Breast irradiation Plus simultaneous tumor bed Boost — hypo-fractionated irradiation for experimental group and normal fractionated irradiation for comprator group

SUMMARY:
In this study,the eligible breast cancer patients will be randomized divided into two groups. the study group receive the accelerated hypo-fractioned whole breast irradiation with a concurrent boost to the tumor bed (WBI 2.5Gy x18 and SIB 2.88Gy x18) and the control group receive conventional fractioned whole breast irradiation with a concurrent boost to the tumor bed(WBI 1.8Gy x28 and SIB 2.15Gy x28). All radiotherapy will be delivered by external beam-intensity modulated radiotherapy. the purpose of this study is to assess whether the accelerated hypo-fractioned is non-inferior to the conventional fractionated radiotherapy. The outcomes evaluation will include acute toxicity , late toxicity including breast fibrosis and cardiac disease, cosmetic outcome ,local control and survival outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients has had breast conserving surgery
2. age ≥ 18 and ≤ 65 years
3. with a histological diagnosis of invasive carcinoma of the breast
4. with pathological stage of T1-2N0-1M0
5. multidisciplinary decision of adjuvant WBI with a boost to the tumor bed
6. informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

1. patients treated with Mastectomy
2. Need for lymph node irradiation
3. positive or close(≤ 1 mm) surgical margin
4. treated with neoadjuvant chemotherapy before surgery
5. Bilateral malignancy of the breast (synchronous or metachronous)
6. Pregnant or breastfeeding
7. Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
8. Patient unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Degree of acute skin toxicity | 2 Weeks after the end of radiotherapy.
  To determine the acute toxicity of accelerated hypo-fractionated whole breast irradiation with concurrent boost to the tumor bed in 18 fractions and whether it will be non-inferior to the conventional fractionated WBI with a concurrent boost

SECONDARY OUTCOMES:
local control | From data of randomization until 60 months after the end of radiotherapy of last patients
  To determine the local control in women with early stage breast cancer treated with accelerated hypo-fractionated whole breast irradiation with concurrent boost to the tumor bed in 18 fractions and whether it will be non-inferior to the conventional fractionated WBI with a concurrent boost
Degree of chronic skin toxicity and cosmesis after radiotherapy | 6 months after radiotherapy
  To assess the chronic skin toxicity and measure cosmesis using the Harvard cosmoses scale in patients and to determine whether the accelerated hypo-fractionated WBI with a concurrent boost is non-inferior to standard WBI with concurrent boost.
Degree of chronic skin toxicity and cosmesis after radiotherapy | 2 years after radiotherapy
  To assess the chronic skin toxicity and measure cosmesis using the Harvard cosmoses scale in patients and to determine whether the accelerated hypo-fractionated WBI with a concurrent boost is non-inferior to standard WBI with concurrent boost.
Degree of chronic skin toxicity and cosmesis after radiotherapy | 5 years after radiotherapy
  To assess the chronic skin toxicity and measure cosmesis using the Harvard cosmoses scale in patients and to determine whether the accelerated hypo-fractionated WBI with a concurrent boost is non-inferior to standard WBI with concurrent boost.
overall survival | From date of randomization until 60 months after the end of radiotherapy of last patients
  To determine whether the overall survival after hypo-fractionated breast radiation with concurrent boost is non-inferior to conventional fractionated radiation therapy with concurrent boost.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiyan Road No.440, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided